CLINICAL TRIAL: NCT03656432
Title: Effect of CPP-ACP Pastes With/Without Fluoride on White Spot Lesion Progression, Salivary pH and Fluoride Release in High Caries Risk Patients A Randomized Clinical Trial
Brief Title: Effect of CPP-ACP With/Without Fl on White Spot Lesion,Salivary pH and fl Release in High Caries Risk Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Doaa Gamal, Principal Investigator and PHD student at Conservative Dentistry Department, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CEBD-CU-2018-08-29
Record Dates: First submitted 2018-08-30; First posted 2018-09-04 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Caries
Keywords: CPP-ACP pastes; CPP_ACPF; Fluoride release; early carious lesion
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CPP-ACP paste (Experimental): MI Paste represents an alternative remineralizing agent that prevents the early demineralization, it is capable of stabilizing calcium phosphate, maintaining the supersaturation of these ions in the oral environment by binding with them and transport them in the form of amorphous calcium phosphate. They can enhance remineralization, decrease demineralization or even both in an acid challenge to teeth surfaces.
  Interventions: Drug: CPP-ACP paste
- CPP-ACP containing fluoride (Experimental): MI paste plus contains fluoride 0.2% (900 ppm) that is very similar to the amount of fluoride in the toothpaste binds to the tooth surfaces and plaque and provides biocompatible calcium, phosphate and fluoride in a localized way. So, it provides all the ions needed to build fluorapatite crystals that are more resistant to the acid attack compared to hydroxyapatite
  Interventions: Drug: CPP-ACP paste
- toothpaste contains fluoride (Active Comparator): Fluoridated Toothpaste are the most significant and worldwide spread forms of caries control used globally as the greater acceptability of toothpaste makes its regular use more likely, thereby improving effectiveness
  Interventions: Drug: CPP-ACP paste

INTERVENTIONS:
Drug: CPP-ACP paste — The complex CPP-ACP derived from a milk protein called casein. CPP-ACP represents an alternative remineralizing agent that prevents the early demineralization, it is capable of stabilizing calcium phosphate, maintaining the supersaturation of these ions in the oral environment by binding with them and transport them in the form of amorphous calcium phosphate. They can enhance remineralization, decrease demineralization or even both in an acid challenge to teeth surfaces.
  Other Names: CPP-ACP containing fluoride paste

SUMMARY:
Effect of CPP-ACP pastes with/without Fluoride on White spot lesion progression, salivary pH and fluoride release in high caries risk Patients, over 3 month period using VistaCam, Digital pH meter and Selective ion electrode.

DETAILED DESCRIPTION:
Dental caries is the most prevalent disease affecting the Human beings, it is a complex disease affecting teeth, which is caused by imbalance between demineralization and remineralization process in the oral cavity.

Preventive measures will stop the development of early caries lesions or even will direct the progression of this early carious lesions towards remineralization.

Nowadays, researchers have focused on non-invasive techniques to prevent early caries lesions appearance. In recent years, a calcium and phosphate remineralization technology has been introduced to decrease their incidence that relies on Casein Phospho-Peptide-Amorphous Calcium Phosphate (CPP-ACP).

The complex CPP-ACP derived from a milk protein called casein. CPP-ACP represents an alternative remineralizing agent that prevents the early demineralization, it is capable of stabilizing calcium phosphate, maintaining the supersaturation of these ions in the oral environment by binding with them and transport them in the form of amorphous calcium phosphate. They can enhance remineralization, decrease demineralization or even both in an acid challenge to teeth surfaces.

CPP-ACP with sodium fluoride 0.2% (900 ppm) that is very similar to the amount of fluoride in the toothpaste binds to the tooth surfaces and plaque and provides biocompatible calcium, phosphate and fluoride in a localized way. So, it provides all the ions needed to build fluorapatite crystals that are more resistant to the acid attack compared to hydroxyapatite . It also has a preventive role in the pH control as it might be able to improve pH levels in different areas in the oral cavity.

Early enamel demineralization is frequently observed as white spot lesions (WSLs) which are opaque enamel areas created by mineral loss from the subsurface layer of enamel. These areas are also defined as incipient or enamel caries. WSLs are the precursors for caries cavities and their milky color may cause esthetic problems .

Taking into consideration that caries detection by eyesight is better for cavitated lesions than for non-cavitated early lesions. Moreover, the visual examination is a subjective method and so it has a lower reproducibility in detecting occlusal caries. Also, radiographic examination has shown high specificity and poor sensitivity for non-cavitated lesions, underestimating the lesion depth . Therefore, the detection of these early carious lesions (WSL) in the initial stage with optimum efficiency achieved by a variety of technologies one of them is the use of autofluorescence technique (VistaCam) for the early detection and diagnosis of these 8 incipient lesions . Studies have shown that white spot lesions can take only one month to develop .

The VistaCam is an intraoral fluorescence camera that illuminates teeth with a violet light (405 nm) and captures the reflected light as a digital image. Which is then is filtered contains the green yellow fluorescence of normal teeth with a peak at 510 nm, as well as the red fluorescence of bacterial metabolites with a peak at 680 nm. The software quantifies the green and red fluorescent light on a scale from 0 to 3 as a ratio of red to green, showing the areas with a higher than healthy tooth ratio .

Although promising, investigations dealing with the effect of CPP-ACP products on plaque and salivary pH levels and in the high caries risk patient appear to be limited and have not been conducted in the form of randomized clinical trials.

Therefore, the purpose of this study was to evaluate the effects of recommending a CPP-ACPF product on salivary pH levels and measuring the amount of fluoride remains in the saliva after using it in high caries risk patients, and also monitoring the prevention of new white spot lesions during the use of CPP_ACP with and without fluoride by using the vistaCam as a randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Age range from 17-30 years
* Males or females
* High caries risk patients defined according to American Dental Association (ADA)
* Systematically healthy
* Not taking any medication interfering with saliva secretion
* Co-operative patients approving to participate in the trial
* signed informed consent

Exclusion Criteria:

* Patients younger than 17 years old or older than 30 years old.
* Disabilities
* Subjects suffering from any medical or systematic disease
* Smokers
* Pregnant females
* Allergy to milk derivatives.
* using any other agents containing fluoride
* presence of untreated caries lesions.

Ages: 17 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 42 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
White Spot Lesion (WSL) progression | (T1) baseline before application, (T2) immediate after application, (T3) 1 day, (T4) 1 week and (T5) 1 month.
  The researcher will inspect the development of any new WSLs in the oral cavity in the clinic of Conservative Dentistry Department Cairo University. The software quantifies the green and red fluorescent light on a scale from 0 to 3 as a ratio of red to green, showing the areas with a higher than healthy tooth ratio.

SECONDARY OUTCOMES:
unstimulated Salivary pH change | (T1) baseline before application, (T2) immediate after application, (T3) 1 day, (T4) 1 week and (T5) 1 month.
  The researcher will collect unstimulated saliva pH samples from outpatient clinic at Conservative Dentistry Department Cairo University which will be measured immediately using digital pH meter. It has no measuring unit, but it only displays numerical value.
stimulated Fluoride Release | For the WSLs assessment, (T1) baseline before application, (T2) 1 month and (T3) 3 months
  The researcher will collect stimulated salivary sample from the participant for fluoride release measurement by selective ion electrode in ppm(mg/l).

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed R Farid, PhD, Study Director — Professor of Conservative Dentistry, Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Poureslami H, Hoseinifar R, Khazaeli P, Hoseinifar R, Sharifi H, Poureslami P. Changes in the Concentration of Ions in Saliva and Dental Plaque after Application of CPP-ACP with and without Fluoride among 6-9 Year Old Children. J Dent Biomater. 2017 Mar;4(1):361-366. PMID 28959766
- [Background] Sinfiteli PP, Coutinho TCL, Oliveira PRA, Vasques WF, Azevedo LM, Pereira AMB, Tostes MA. Effect of fluoride dentifrice and casein phosphopeptide-amorphous calcium phosphate cream with and without fluoride in preventing enamel demineralization in a pH cyclic study. J Appl Oral Sci. 2017 Nov-Dec;25(6):604-611. doi: 10.1590/1678-7757-2016-0559. PMID 29211281
- [Background] Heshmat H, Banava S, Mohammadi E, Kharazifard MJ, Mojtahedzadeh F. The effect of recommending a CPP-ACPF product on salivary and plaque pH levels in orthodontic patients: a randomized cross-over clinical trial. Acta Odontol Scand. 2014 Nov;72(8):903-7. doi: 10.3109/00016357.2014.920515. Epub 2014 May 26. PMID 24856191
- [Background] Ebrahimi M, Mehrabkhani M, Ahrari F, Parisay I, Jahantigh M. The effects of three remineralizing agents on regression of white spot lesions in children: A two-week, single-blind, randomized clinical trial. J Clin Exp Dent. 2017 May 1;9(5):e641-e648. doi: 10.4317/jced.53582. eCollection 2017 May. PMID 28512540
- [Background] Tassery H, Levallois B, Terrer E, Manton DJ, Otsuki M, Koubi S, Gugnani N, Panayotov I, Jacquot B, Cuisinier F, Rechmann P. Use of new minimum intervention dentistry technologies in caries management. Aust Dent J. 2013 Jun;58 Suppl 1:40-59. doi: 10.1111/adj.12049. PMID 23721337
- See also: Topical Tooth Créme Containing Calcium, Phosphate & Fluoride — http://www.gcamerica.com/products/preventive/MI_Paste/index.php